CLINICAL TRIAL: NCT04923763
Title: The Establishment of Tongue Examination Analysis From the Video Recording
Status: Recruiting | Type: Observational
Sponsor: China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Han-Kuei Wu, Assistant Professor, China Medical University, Taiwan
Other Study IDs: Tongue_VA
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Medicine, Chinese Traditional
Keywords: tongue examination; video recording; artificial intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tongue_examination: The general public will be invited for tongue examination. The data will be used to establish the automatic tongue video analysis system.

SUMMARY:
This project intends to record the process of tongue extension through a dynamic video, and establish the tongue examination analysis from the video recording.

In this study, 300 general public will be invited for examinations, and high-quality tongue examination videos will be recorded by digital cameras. After the tongue examination video is properly calibrated, the computer analyzes the tongue examination parameters of each frame and the dynamic parameters, thereby establishing the automatic tongue video analysis system

DETAILED DESCRIPTION:
Traditional Chinese medicine (TCM) doctors use tongue examination to investigate the distribution of qi and blood in the human body and the changes in cold and heat, deficiency and excess. This is a characteristic diagnosis of Chinese medicine and is rich in important clinical diagnostic information. In recent years, tongue examination through computer image analysis has been a fairly mature technology, but its application still has many limitations. A proper tongue examination image capture must be performed by a well-training staff, and errors caused by the operator cannot be avoided. These restrictions are not conducive to the popularization of tongue examination applications. This project intends to record the process of tongue extension through a dynamic video, and establish the tongue examination analysis from the video recording.

In this study, it is estimated that 300 subjects will be admitted to the China Medical University and its cooperative medical facilities. The general public will be invited for examinations, and high-quality tongue examination videos will be recorded by digital cameras. After the tongue examination video is properly calibrated, the computer analyzes the tongue examination parameters of each frame and the dynamic parameters, thereby establishing the automatic tongue video analysis system.

This study is different from recording the tongue with photos in the past, but uses dynamic movies to record the tongue extension process, avoiding the influence of external light source and tongue placement, seeking the best timing for tongue diagnosis, and it is expected to produce automatic dynamic video tongue examination analysis, as an innovative analysis model of TCM tongue examination. Results are expected to reduce operating errors and promote the popularization of automated tongue examination analysis. In the future, it may be applied to mobile phones or wearable devices to improve the practicality of TCM tongue examination in telemedicine and the personalized medicine.

ELIGIBILITY:
Inclusion Criteria:

* general public

Exclusion Criteria:

* unable to complete tongue examination

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Convenience sampling in the China Medical University and its cooperative medical facilities.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tongue video analysis | one day
  The general public will be invited for tongue examination with video record. The data will be used to establish the automatic tongue video analysis system.

SECONDARY OUTCOMES:
Heart rate variability | one day
  Heart rate variability will be evaluated by "Wegene" Handheld ECG Monitor (8Z11) to investigate the possible correlation with tongue video analysis parameters.
Chinese medicine constitution | one day
  Chinese medicine constitution will be evaluated by the Constitution Tendency Questionnaire (CTQ) investigate the possible correlation with tongue video analysis parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hung Tien, Bachelor, Study Director — China Medical University, Taiwan
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided